CLINICAL TRIAL: NCT07168070
Title: Effects of Individualized Physical Therapy and Group Physical Therapy on Functional Outcomes in Patients With Femoral Neck Fracture in Gaza Strip
Acronym: neck of femure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University - Gaza (Other)
Responsible Party: Principal Investigator, Mohammed Nabil Matar, clinical instructor and researchs coordinator, Al-Azhar University - Gaza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20220033; 232855 (Other: Ministry of Health - Palestine)
Record Dates: First submitted 2025-08-20; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Orthopaedic Disorders; Neck of Femur Fracture
Keywords: NoF
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Physical Therapy Modalities; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized Physical Therapy Program (Experimental): Participants will receive one-on-one physiotherapy sessions, 45 minutes each, three times per week for 8 weeks, including range of motion, strengthening, balance, and gait training.
  Interventions: Other: physical therapy and exercise; Behavioral: group physical therapy vs individualized physical therapy; Other: Group Physical therapy
- group physical therapy (Experimental): group of people given the same treatment at the time
  Interventions: Other: physical therapy and exercise; Behavioral: group physical therapy vs individualized physical therapy; Other: Group Physical therapy

INTERVENTIONS:
Other: physical therapy and exercise — Participants will receive one-on-one physiotherapy sessions, 45 minutes each, three times per week for 6 weeks. Sessions will include range of motion, strengthening, balance, and gait training.
  Home-based Exercise Participants will be instructed to perform a structured home exercise program to complement in-clinic sessions.
  Other Names: One person-focused physical therapy session
Behavioral: group physical therapy vs individualized physical therapy — group physical therapy vs individualized physical therapy
Other: Group Physical therapy — Participants will attend group physiotherapy sessions, where several patients receive treatment at the same time. Each session lasts 45 minutes, three times per week for 6 weeks, and includes range of motion, strengthening, balance, and gait training.
  Other Names: Group physical therapy vs individualized physical therapy

SUMMARY:
The research explores how individualized, one-on-one physical therapy programs versus group-based therapy sessions influence recovery in terms of functional mobility, pain reduction, muscle strength, balance, and overall quality of life. Patients were recruited from healthcare facilities in the Gaza Strip and were randomly assigned to either intervention group.

1.2 Justification of the study This study provides important evidence on the role of group Physical Therapy in rehabilitation outcomes, which is a key factor in enhancing both the physical and psychological recovery of patients with femoral neck fractures. By focusing on the impact of rehabilitation environments, particularly the comparison between individualized Physical Therapy and group Physical Therapy, this research addresses a critical gap in the existing literature. While much of the current research has concentrated on the physical aspects of recovery, the influence of social engagement and environmental factors remains underexplored, despite their potential to significantly improve outcomes. The findings of this study may help to inform clinical guidelines by providing a clearer understanding of how group-based rehabilitation, which encourages social interaction, could be integrated into recovery protocols for better results. Additionally, the insights gained from this research have the potential to guide policymakers and healthcare providers in the development of more effective rehabilitation programs tailored to the specific needs of patients. By optimizing rehabilitation strategies based on the rehabilitation environment, this study aims to enhance recovery times and overall Functional independency in ADLs for patients, ultimately leading to better health outcomes and a more efficient use of healthcare resources.

1.3 Study objectives 1.3.1 General objective To evaluate the effect of a tailored exercise intervention program on patients' QoL among patients who have undergone lumbar discectomy.

1.3.2 Specific objectives

1. To examine the effect of tailored exercise intervention in reducing pain among patients who have undergone lumbar discectomy.
2. To investigate the effect of a tailored exercise intervention program in reducing the level of disability among patients who have undergone lumbar discectomy.
3. To assess the effect of a tailored exercise intervention program in reducing the level of depression and anxiety among patients who have undergone lumbar discectomy.

1.4 Hypothesis To compare the effects of individualized Physical Therapy and group Physical Therapy on functional outcomes in patients with femoral neck fractures in Gaza strip.

1.5 Specific Objectives

To evaluate the effects of individualized Physical Therapy Program on functional independence in the ADLs, sleep quality, depression and anxiety in patients with femoral neck fractures in Gaza strip.

To evaluate the effects of group Physical Therapy Program on functional independence in the ADLs, sleep quality, depression and anxiety in patients with femoral neck fractures in Gaza Strip.

1.6. Hypothesis 1.6.1 H0 There will be no significant difference in functional independence in ADLs between patients recovering from femoral neck fractures who undergo rehabilitation in individualized Physical Therapy and group Physical Therapy.

1.6.2 H1 There will be a significant difference in functional independence in ADLs between patients recovering from femoral neck fractures who undergo rehabilitation in individualized Physical Therapy and group Physical Therapy.

There will be a significant difference in sleep quality between patients recovering from femoral neck fractures who undergo rehabilitation in individualized Physical Therapy and group Physical Therapy.

There will be a significant difference in depression and anxiety symptoms between patients recovering from femoral neck fractures who undergo rehabilitation in individualized Physical Therapy and group Physical Therapy.

1.7 Research Questions

Is there a significant difference in functional independence in ADLs between patients recovering from femoral neck fractures who undergo rehabilitation in individualized Physical Therapy and group Physical Therapy? Is there a significant difference in sleep quality between patients recovering from femoral neck fractures who undergo rehabilitation in individualized Physical Therapy and group Physical Therapy? Is there a significant difference in depression and anxiety symptoms between patients recovering from femoral neck fractures who undergo rehabilitation in individualized Physical Therapy and group Physical Therapy? What are the baseline levels of functional independence in ADLs, depression, anxiety, functional mobility, and sleep quality among patients with femoral neck fractures screened for the study?

DETAILED DESCRIPTION:
Femoral neck fractures are a significant public health concern, particularly among the elderly population. According to Dyer the incidence of hip fractures is rising, leading to a marked decline in physical function and increased morbidity and mortality rates . For patients experiencing hip fractures, key outcomes such as survivability, morbidity, and functional independence in activities of daily living (ADLs) are profoundly impacted. Hip fractures abruptly alter a person's life and may increase their reliance on others to carry out everyday tasks.

Femoral neck fractures have a significant negative impact on quality of life by creating mobility issues. After being hospitalized for a hip fracture, only roughly 60% of patients are able to walk normally again. A growing percentage of people who survive neck of fracture injuries go on to suffer from varying degrees of later handicap, such as the development of excruciating osteoarthritis in their hip joints, a high risk of falls, and additional hip fracture injuries. Furthermore, Fractured individuals experience lower quality of life due to poor balance and movement, as well as reduced functional and social independence. This suggests that many people never resume their pre-fracture way of life.

While much of the existing research has focused on the physical aspects of recovery, such as restoring pre-fracture functional abilities, less attention has been given to the psychological factors that influence functional mobility. Successful recovery is not solely dependent on physical rehabilitation but also on psychological well-being. Psychological comorbidities are significantly associated with both mortality and functional outcome in patients with neck of femur fractures. More than half of all patients reported continued sleep disturbance 3 months post orthopaedic operation. Early identification and management of sleep disturbances can improve functional and emotional recovery outcomes. Fatigue from poor sleep may hinder adherence to home exercise regimens, impacting overall recovery .

Also, patients with a femoral neck fracture are at an increased risk of subsequent major depression. Interestingly, patients undergoing surgery for femoral neck fracture with comorbid psychological problems are at increased risk for non-routine discharge. These problems are independently associated with an increased risk for post-operative complications. An awareness of these risks should optimize preoperative multidisciplinary patient care planning so as to maximize patient outcome.

In patients with a hip fracture, post-operative rehabilitation can enhance clinical results and quality of life. Prolonged immobilization can lead to functional decline and complications like falls and pressure ulcers. Early mobilization helps prevent these issues. A systematic review conducted by Peeters, et al found that home-based rehabilitation programs incorporating strength exercises significantly improved health status components. Additionally, stone et al. found that a more intensive community-based multimodal therapy (six or more in-person sessions per week) did not lead to better outcomes at three months compared to a less frequent regimen (three or fewer sessions per week).

Group-based rehabilitation strategies have also been shown to enhance functional outcomes. Coulter found that group Physical Therapy following joint replacement surgery yielded functional recovery results comparable to customized home-based physical therapy. Similarly, Tarakci demonstrated that supervised group exercise training significantly improved balance and functional status in patients with multiple sclerosis, further reinforcing the effectiveness of group-based interventions. On the other hand, O'Keeffe compared the efficacy of individual and group Physical Therapy exercise programs for musculoskeletal problems. Their findings revealed no clinically significant differences between the two approaches in terms of pain and impairment outcome. Previous research suggests that group engagement during rehabilitation can enhance motivation and improve recovery outcomes. In contrast, individualized rehabilitation may provide more focused care but could lack the psychological and social benefits associated with group-based therapy. So, it is not clear whether exercises performed in a group or individualized settings are better for improving outcomes post femoral neck fractures.

There is a gap in the literature regarding the impact of rehabilitation environments (group and individualized setting) on functional mobility and ADL independence in patients recovering from femoral neck fractures. To our knowledge, a few studies have examined the influence of Physical Therapy interventions on functional and psychological factors in this population. Thus, this study aims to bridge this gap by exploring the effect of different rehabilitation settings on functional mobility, ADL independence, sleep and psychological factors in patients recovering from femoral neck fractures.

Statement of The Problem

Despite the profound effects of femoral neck fractures on both physical and mental health, there is a notable lack of comprehensive rehabilitation protocols tailored to address the multifaceted needs of these patients. Current rehabilitation practices often focus primarily on physical recovery, neglecting the critical psychological and sleep-related aspects that are essential for holistic recovery. Femoral neck fractures often lead to a decline in physical function, resulting in increased dependence on caregivers and a reduced ability to perform activities of daily living (ADLs). Furthermore, the aftermath of femoral neck fractures is frequently accompanied by sleep disturbances, which can exacerbate fatigue and hinder recovery. The psychological ramifications are equally concerning, as many patients experience heightened levels of depression and anxiety following their injury, further complicating their rehabilitation process Study objectives

General objective:

To compare the effects of individualized Physical Therapy and group Physical Therapy on functional outcomes in patients with femoral neck fractures in Gaza strip.

Specific Objectives:

To evaluate the effects of individualized Physical Therapy Program on functional independence in the ADLs, sleep quality, depression and anxiety in patients with femoral neck fractures in Gaza strip.

To evaluate the effects of group Physical Therapy Program on functional independence in the ADLs, sleep quality, depression and anxiety in patients with femoral neck fractures in Gaza Strip.

Hypothesis H0 There will be no significant difference in functional independence in ADLs between patients recovering from femoral neck fractures who undergo rehabilitation in individualized Physical Therapy and group Physical Therapy.

H1 There will be a significant difference in functional independence in ADLs between patients recovering from femoral neck fractures who undergo rehabilitation in individualized Physical Therapy and group Physical Therapy.

There will be a significant difference in sleep quality between patients recovering from femoral neck fractures who undergo rehabilitation in individualized Physical Therapy and group Physical Therapy.

There will be a significant difference in depression and anxiety symptoms between patients recovering from femoral neck fractures who undergo rehabilitation in individualized Physical Therapy and group Physical Therapy.

1.7 Research Questions

Is there a significant difference in functional independence in ADLs between patients recovering from femoral neck fractures who undergo rehabilitation in individualized Physical Therapy and group Physical Therapy? Is there a significant difference in sleep quality between patients recovering from femoral neck fractures who undergo rehabilitation in individualized Physical Therapy and group Physical Therapy? Is there a significant difference in depression and anxiety symptoms between patients recovering from femoral neck fractures who undergo rehabilitation in individualized physical therapy and group physical therapy? What are the baseline levels of functional independence in ADLs, depression, anxiety, functional mobility, and sleep quality among patients with femoral neck fractures screened for the study? 1.5 Theoretical and Operational Definition of Terms Femoral neck fractures occur in the femoral neck, which is where the femoral head and shaft meet. Because of its placement, the femoral neck is prone to fracture, and in cases where it is displaced, disruption of the femoral head's blood supply is a major issue.

Group physical therapy is a rehabilitation technique in which a professional physical therapist supervises therapeutic exercises or activities for two or more patients at the same time with the purpose of safely and effectively addressing individual or shared goals Individualized Physical Therapy is a rehabilitation technique in which a professional physical therapist supervises therapeutic exercises or activities for only one patient

ELIGIBILITY:
Inclusion Criteria:

* Patients Male and female aged 50 years or older.
* Diagnosed with unilateral femoral neck fracture and underwent surgical treatment.

Exclusion Criteria:

* Patients with bilateral fractures or multiple trauma injuries.
* Patients with pathological related fractures.
* Presence of severe cognitive impairment (e.g., advanced dementia).
* Severe neurological disorders (e.g., stroke, Parkinson's disease) that affect mobility.
* Unstable cardiovascular conditions that limit exercise participation.
* Not willing to provide informed consent.
* Unable to participate in Physical Therapy with or without assistance

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-22 (Estimated); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-10-21 (Estimated)

PRIMARY OUTCOMES:
Barthel Index | 6 weeks
  a tool used to evaluate the functional independence in ADLs (toileting, bathing, eating, dressing, continence, transfers, and ambulation). Each task received a numerical score based on whether the patient required physical assistance to perform it. A patient scoring 0 points would be dependent in all assessed ADLs, whereas a score of 100 would reflect independence in all activities. Barthel Index is a valid and reliable tool to measure the functional independence. It has adequate reliability (intraclass correlation coefficient ≥ 0.962) and internal consistency (Cronbach's alpha = 0.942)
Hospital Anxiety and Depression Scale (HADS) | 6 weeks
  Hospital Anxiety and Depression Scale (HADS) is a self-assessment tool used to screen for anxiety and depression in patients, especially in non-psychiatric medical settings. It consists of 14 items: 7 for anxiety (HADS-A) and 7 for depression (HADS-D), each scored on a 4-point scale (0-3). Scores range from 0-21 for each subscale, with higher scores indicating more severe symptoms
Subjective sleep quality | 6 weeks
  Sleep quality will be assessed by Pittsburgh Sleep Quality Index (PSQI). PSQI consists of 19-items that assess seven dimensions: duration of sleep, subjective sleep quality, sleep latency, sleep disturbance, habitual sleep efficiency, taking sleep medications, and daytime dysfunction over the last month. Cronbach's α for the seven component scores that comprise the PSQI global score was 0.74, which suggests good internal consistency.

IPD SHARING:
Plan to Share IPD: Yes
The de-identified individual participant data (IPD) underlying the results of this study will be made available to other researchers upon reasonable request. Data to be shared include demographic information, baseline characteristics, and outcome measures related to functional recovery, mobility, and quality of life following femoral neck fracture.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available within 6 months after publication of the primary results and will remain accessible for 5 years thereafter.
Access Criteria: Researchers who provide a methodologically sound proposal and obtain approval from a relevant ethics committee will be granted access. Requests should be directed to the principal investigator via email. The data will be shared in de-identified form only, to ensure patient confidentiality, and solely for academic and research purposes.